CLINICAL TRIAL: NCT05056324
Title: Internet-based Vestibular Rehabilitation Versus Standard Care After Acute Onset Vertigo
Brief Title: Web-based Rehab After Acute Vertigo
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Umeå University (Other)
Collaborators: University Hospital, Umeå (Other); Sundsvall Hospital (Other); Sahlgrenska University Hospital (Other); Västernorrland County Council, Sweden (Other Government); Södra Älvsborg Hospital (Other); Karolinska University Hospital (Other); University Hospital, Linkoeping (Other); Sunderby Hospital (Other); Capio Sankt Görans Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Web-based vertigo rehab; CIV-21-05-036744 (Other: Swedish Medical Products Agency)
Record Dates: First submitted 2021-09-07; First posted 2021-09-24 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2024-08

CONDITIONS: Acute Vestibular Syndrome
Keywords: acute vestibular syndrome; vertigo; vestibular rehabilitation
MeSH Terms: conditions — Vertigo | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention group (Experimental)
  Interventions: Device: Online vestibular rehabilitation tool
- Control group (Active Comparator)
  Interventions: Other: Standard care (written instructions leaflet)

INTERVENTIONS:
Device: Online vestibular rehabilitation tool — For those randomized to the intervention group, a 6 weeks duration vestibular rehabilitation will be delivered using an online tool (YrselTräning)
  Arms: Intervention group
Other: Standard care (written instructions leaflet) — For those randomized to the control group, a 6 weeks duration standard vestibular rehabilitation will be delivered using a written instructions leaflet
  Arms: Control group

SUMMARY:
Acute onset vertigo is common and entails much suffering with persisting symptoms at 3 months after onset in up to half of those afflicted. Vestibular rehabilitation to aid recovery is not readily available. The purpose of this study is to investigate the effects on vertigo symptoms of a 6-week online vestibular rehabilitation tool compared with standard care (written instructions leaflet) after acute onset vertigo.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years old; and
* The subject has given written consent to participate in the study; and
* New acute onset dizziness or vertigo since ≥24 hours with pathological spontaneous or gaze-evoked nystagmus (i.e. an acute vestibular syndrome, AVS). The nystagmus as described above must be present at investigation between 24 hours and 7 days from onset, spontaneously, gaze-evoked or head-shake evoked and documented; and
* Screening and inclusion within 7 days of onset of continuous symptoms; and
* Symptomatic at inclusion

Exclusion Criteria:

* Pre-existing vestibular disease or neurological disease anticipated to affect the ability to participate in the study or the effect of the intervention. N.B: Recurring AVS with no set diagnosis before inclusion is accepted, as is past transient neurological diseases such as TIA or migraine; or
* Inability to use the online rehabilitation tool, e.g. due to not having access to a computer, tablet or smartphone, not having access to the internet or lacking in experience with such tools; or
* Mental inability, reluctance or language difficulties that result in difficulty understanding the meaning of study participation; or
* Medical and/or physical contraindications to making the required head movements (e.g. vertebral dissection) or otherwise participating in the training and testing exercises or data collection; or
* Medication or other substance intake which can affect the ability to participate in the study or the reliability of the measurement methods. These medications include regular use of: Anticonvulsants, antiemetics/motion sickness medications, benzodiazepines, neuroleptics. Transient corticosteroid and/or antiemetic treatment related to the current vertigo is accepted.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 184 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2024-02-01 (Actual); Study Completion 2025-03-12 (Actual)

PRIMARY OUTCOMES:
The between group mean Vertigo Symptom Scale Short Form (VSS-SF) score difference | 6 weeks after vertigo onset
  VSS-SF uses a five-point Likert scale: 0 (never), 1 (a few times), 2 (several times), 3 (quite often [every week]), and 4 (very often [most days]). The score ranges from 0 to 60. A higher score indicates worse symptoms.

SECONDARY OUTCOMES:
The between groups mean Dizziness Handicap Inventory (DHI) score | 6 weeks and 3 months after vertigo onset
  The Dizziness Handicap Inventory (DHI) uses a three-point scale to rate each item: 0 (no), 2 (sometimes), and 4 (always). The score ranges from 0 to 100. A higher overall score indicates more severe handicap.
The between groups changes in timed 25-foot walk test (T25-FW)); body sway during standing and walking; and the mobility | From baseline to 6 weeks and 3 months
The between groups changes in video head impulse test (vHIT, site-dependent) | 6 weeks and 3 months after vertigo onset
The between groups changes in video head impulse test (vHIT, site-dependent) measured lateral canal VOR gain and saccades | From baseline to 6 weeks and 3 months
The between groups mean vertigo symptom scale short form (VSS-SF) score | 12 months after vertigo onset
  VSS-SF uses a five-point Likert scale: 0 (never), 1 (a few times), 2 (several times), 3 (quite often [every week]), and 4 (very often [most days]). The score ranges from 0 to 60. A higher score indicates worse symptoms.
The between group pedometer-derived mean weekly number of steps walked since last visit | 3 months after vertigo onset
The between groups mean number of weekly training sessions | 6 weeks after vertigo onset
Register-based search for health economic effects on all levels of care (primary, specialized) and society (sick leave) | 12 months
The difference in kinematic output between measurement systems (i.e., multi-sensor and mobile app) | Three months after symptom onset
The reliability of the Swedish VSS-SF translation | Six weeks after symptom onset
The frequency of BPPV at 6 weeks and 3 months after AVS onset using a BPPV specific questionnaire and positional nystagmus tests | 6 weeks and 3 months after vertigo onset

OTHER OUTCOMES:
The proportion of participants who has experienced falls/fractures since study start | 6 weeks, 3 months and 12 months
The number of falls/fractures in each study arm | 6 weeks, 3 months and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Jonatan Salzer, MD, PhD, Principal Investigator — Umeå University
Locations (9):
- Sweden (9):
  - Södra Älvsborg Hospital, Borås
  - Sahlgrenska University Hospital, Gothenburg
  - University Hospital Linköping, Linköping
  - Sollefteå Hospital, Sollefteå
  - Sunderby Hospital, Södra Sunderbyn
  - Capio Sankt Görans Hospital, Stockholm
  - Karolinska University Hospital, Stockholm
  - Sundsvall Hospital, Sundsvall
  - University Hospital Umeå, Umeå

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Surano S, Faergemann E, Granasen G, Salzer J. The reliability and validity of the Swedish translation of the Vertigo Symptom Scale - short form in a cohort with acute vestibular syndrome. Ann Med. 2025 Dec;57(1):2457517. doi: 10.1080/07853890.2025.2457517. Epub 2025 Feb 10. PMID 39928092
- [Background] Surano S, Grip H, Ohberg F, Karlsson M, Faergemann E, Bjurman M, Davidsson H, Ledin T, Lindell E, Mathe J, Tjernstrom F, Tomanovic T, Granasen G, Salzer J. Internet-based vestibular rehabilitation versus standard care after acute onset vertigo: a study protocol for a randomized controlled trial. Trials. 2022 Jun 16;23(1):496. doi: 10.1186/s13063-022-06460-0. PMID 35710448